CLINICAL TRIAL: NCT05242627
Title: Development, Implementation, and Evaluation of a Firearm-Safety Counseling Educational Module for Medical Students
Brief Title: Firearm-Safety Counseling: Medical Student Training
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Gary Holland, MD, Distinguished Professor of Ophthalmology, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-000968
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Medical Student Firearm Epidemiology Knowledge; Medical Student Firearm Safety Knowledge; Medical Student Initiated Clinical Firearm Safety Counseling
Keywords: Firearm; Firearm Safety Counseling; Suicide Prevention; Medical Education
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Students in the DGSOM Classes of 2023 and 2024 will participate in the same Observed Structured Clinical Exam (OSCE) scenario during their second year of medical school, in which they virtually interview a standardized patient presenting with postpartum depression. The Class of 2023 received no specific training on firearm screening and counseling, while the Class of 2024 participated in an educational module on firearm safety counseling 6-months prior to the OSCE.
Who Masked: Participant
Masking Description: The post-partum OSCE is a regular assessment as part of the DGSOM curriculum. After completing their OSCE, student's will be consented to allow their OSCE to be viewed by the study team (all OSCEs are routinely recorded for assessment purposes) and will be presented with a post-OSCE survey to assess their attitudes and beliefs on firearms as well as their performance on the OSCE. Students in both arms are masked to the fact that their OSCE performance will be evaluated in a comparative study (in addition to evaluation as a part of the standard curriculum) while they are participating in the study. Informed consent for their OSCE to be included in the study will be obtained after the OSCEs have been completed. There will be no prompting about firearms prior to the OSCE. Study results regarding firearm screening and counseling will not factor into the student's grade on the OSCE.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DGSOM Class of 2023 (No Intervention)
- DGSOM Class of 2024 (Experimental)
  Interventions: Behavioral: Clinical Firearm Safety Counseling Module

INTERVENTIONS:
Behavioral: Clinical Firearm Safety Counseling Module — The DGSOM class of 2024 will participate in a mandatory 1-hour module covering four main domains: (1) firearm epidemiology; (2) suicide epidemiology and introduction to "means matter"; (3) firearm counseling; and (4) an example of standardized patient encounter that includes a discussion of firearm safety with the patient. The module will be taught in combination by the study team, subject matter experts, and the DGSOM Standardized Patient Program.
  Arms: DGSOM Class of 2024

SUMMARY:
In the United States, nearly one in every three households contains at least one firearm, and roughly 20-25% of American adults personally own a firearm. Such easy access to firearms is a major contributor to the uniquely high levels of firearm-related violent death in the United States compared with other high-income nations. American physicians are intimately aware of this burden and are positioned to help modify the risks that firearms pose to the health and safety of their patients. Accordingly, it is imperative that physicians learn both how to screen their patients for exposure to firearms and how they can effectively counsel those who are at an increased risk for firearm-related injury on how they might reduce that risk.

Until the 2021-2022 academic year, the David Geffen School of Medicine (DGSOM) at the University of California, Los Angeles (UCLA) did not include in its medical school curriculum a firearm-safety counseling module; the only information pertaining to firearms had been a narrow-in-scope "Clinical Pearl," which gave statistics on the increased risk for fatal injury that firearms pose in the setting of domestic violence. Beginning with the incoming Class of 2025, DGSOM will implement a new curriculum, and the Curriculum Re-design Committee has incorporated a module offering instruction on how to screen for exposure to firearms and counsel patients on firearm-safety. This inclusion follows a pilot module on firearm safety counseling that was presented to the Class of 2023. The current trial will take advantage of these unique circumstances to evaluate the effects of introducing such a module on medical students' attitudes, beliefs, and behaviors related to firearm-safety counseling in the clinical setting. The performance of students in the Class of 2023, who did not receive training, will be compared to that of students in the Class of 2024, who did receive training, during a standardized patient encounter.

The high prevalence of firearms in the US demands that physicians have a working knowledge of how to screen patients for exposure to firearms, and an ability to counsel those who have such exposure on firearm-safety. While physicians believe they should have an active role in screening for risk factors of firearm violence and counsel on firearm safety, experience indicates that they fail to do either routinely. Importantly, physicians cite a lack of training and self-confidence as the major factors preventing them from screening for, and counseling on, firearm safety. A recent study of third-year medical students showed that those who completed a brief (20 minute) module on firearm injury prevention (compared with those who did not) were more likely to report increased self-perceived ability to counsel patients on firearm injury prevention, both immediately and 6 months post intervention; however, the study failed to demonstrate a difference in long-term clinical behavior, suggesting more rigorous training methods are warranted. The investigators hope that educational modules supplemented with simulated patient interactions designed to allow students the opportunity to practice firearm-safety counseling will increase their propensity for engaging in these conversations in the future.

The first innovative aspect of our proposal is that it is introducing an educational module which combines didactic lectures, interactive case-based discussions, and interviews with standardized patients. On a computerized literature search, the investigators found no evidence that such a comprehensive module has been studied. Furthermore, unlike previous studies which have either focused on immediate self-reported confidence or self-reported clinical encounters, the investigators' proposal intends to assess long-term retention of the module content by observing students' clinical practices in an OSCE 6 months after the module is taught. The investigators hypothesize that an educational module will significantly increase both the proportion of second-year medical year students who screen for firearms and the quality of firearm safety counseling.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility Criteria is limited to being a member of the DGSOM Classes of 2023 or 2024.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-10-11 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of firearm screening and counseling in a modified clinical setting. | 1 day
  The prevalence of medical students screening for the presence of firearms and counseling on firearm safety will be assessed during a standardized Observed Structured Clinical Exam (OSCE). The proportion of students who counsel will be reported by the standardized patients and by students who consent to having their OSCE included in the study.

SECONDARY OUTCOMES:
Medical Student's Attitudes and Beliefs on Firearms | Up to 16 months
  Students will complete a survey several months prior to the OSCE on their baseline attitudes and beliefs regarding firearms. Students in the DGSOM Class of 2024 will complete the same survey following the training module.

OTHER OUTCOMES:
Firearm Safety Counseling Quality | 1 day
  The standardized patients, who have been familiarized firearm counseling procedures, will report their subjective view of the quality of the student's counseling. Additionally, the study team will objectively score the counseling based on a predetermined rubric while watching a video of each student-participant's OSCE.

CONTACTS AND LOCATIONS:
Locations (1):
- David Geffen School of Medicine at UCLA, Los Angeles, California, United States